CLINICAL TRIAL: NCT05416294
Title: Neurostimulation an Adjuvant Postoperative Analgesic in Total Knee Replacement (TKR) Surgeries
Acronym: TKR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS014
Record Dates: First submitted 2022-05-26; First posted 2022-06-13 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Arthroplasty, Knee Replacement
Keywords: Knee Replacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Device (Experimental): Participants in this arm will receive an active Primary Relief device placed following the total knee replacement surgery.
  Interventions: Device: Primary Relief
- Placebo Device (Sham Comparator): Participants in this arm will receive an inactive (sham) Primary Relief device placed following the total knee replacement surgery.
  Interventions: Device: Inactive Primary Relief

INTERVENTIONS:
Device: Primary Relief — The group will receive PENS treatment using Primary Relief in addition to the multimodal analgesia (morphine, ketorolac, methyl, prednisolone, adrenaline) including the periarticular infiltration of local anaesthetic and/or femoral or epidural catheter for postoperative pain management (bupivacaine, ropivacaine).
  Arms: Active Device
Device: Inactive Primary Relief — The group will receive a sham device with multimodal analgesia (morphine, ketorolac, methyl, prednisolone, adrenaline), including the periarticular infiltration of local anaesthetic and/or femoral or epidural catheter for postoperative pain management (bupivacaine, ropivacaine).
  Arms: Placebo Device

SUMMARY:
To study and evaluate the effect of using the Primary Relief PENS treatment as adjuvant analgesia for reducing pain in total knee replacement (TKR) patients.

DETAILED DESCRIPTION:
It is a common knowledge that total knee replacement (TKR) surgeries produce great deal of pain in the postoperative period. Superior pain relief is justifiably needed and usually provided. In addition to the conventional methods of pain relief such as continuous epidural block, intrathecal adjuvants, femoral nerve block ± sciatic nerve block, transcutaneous electrical nerve stimulation (TENS) and percutaneous electrical neurostimulation (PENS) have been reported effective by various authors. Recently neurostimulation of auricular nerves via the external auricular surface has shown to alleviate pain after caesarian section. Primary Relief® is percutaneous electrical neuro stimulator designed to administer auricular neurostimulation treatment over 240 hours. Stimulation is performed by sending electrical pulses emitted through needles strategically positioned in the ear. The ear provides numerous points for stimulation within a small area Based on the area of pain relief, chosen points are stimulated. Primary Relief is a miniaturized device designed to administer PENS treatment. Use of this device is recommended for pre-operative, intra-operative and post-operative pain therapy as well as for the treatment of chronic pain.

An advantage over drug therapy is that it avoids the possible side-effects of analgesics and helps in early mobilization following orthopedic surgeries including total knee replacement (TKR), total hip replacement (THR) and shoulder surgeries. Therefore, this study is being undertaken to assess the effect of Primary Relief ® in augmenting pain relief after TKR surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing TKR under regional or general anesthesia and femoral nerve block who consent to participate in the study.

Exclusion Criteria:

* ASA 3 or 4
* Those receiving psychiatric medication
* Those with infection at the site of application.

The following data will be collected

* Intraoperative use of local anesthetics, opioids and other analgesics
* Postoperative details as to the time of application of the device. NPRS in both the groups at multiple intervals, on demand analgesic requirement, overall analgesic consumption during the study period, quality of life questionnaire at the end of the study period and relevant postoperative complications will be noted.
* Rescue analgesics will be considered for breakthrough pain or NPRS > 4. Intravenous Tramadol 50mg will be the first rescue analgesic and if pain is not relieved with Tramadol, opiods will be considered. Non steroidal anti inflammatory drugs will be considered to supplement the above medications if there is no contraindication and if need arises.
* NPRS score will be noted at multiple intervals for 10 days.
* Any nausea, vomiting, giddiness, intolerance to the device will also be noted.
* During the follow up, quality of life questionnaire would be administered and the result noted.

The device will be removed after 10 days of its application. Any redness at the site of application or pain at the site are noted. The study will end with the removal of the device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 0 - 3 days ; 0,2,4,6,8,10,12,18,24,36,48,60,72 hrs from the time of completion of surgery
  To evaluate the pain score in the immediate postoperative period. Pain Score with will be measured on a scale (0 = no pain; 10 = worst imaginable pain).

SECONDARY OUTCOMES:
NPRS Numerical Pain Rating Scale score post-mobilization | 4 - 10 days ; 96,120,144,168,192,216,240 hrs from the time of completion of surgery)
  To evaluate the effect of treatment in reducing the average NPRS scores after mobilization. The measurement will record the daily NPRS scores from day three to ten days.
Total Use of Analgesics and Opioids | OVERALL DOSE IN FIRST 3 DAYS & OVERALL DOSE REQUIRED BETWEEN 4 TO 10 DAYS
  To evaluate the effect of treatment in reducing the overall analgesic and opioid requirement in the immediate postoperative period. The measurement will record the total dose and number of additional analgesics required during the immediate postoperative period at rest.
KOOS Score The Knee injury and Osteoarthritis Outcome Score ( koos) | 5 times planned from 0 - 10 day; (i) 24 hrs before Surgery; (ii) 24 Hrs after completion of surgery; (iii) 72 hrs after completion of Surgery; (iv) 120 hrs after completion of Surgery; (v) At the time of device removal -@240 hrs)
  To assess the effect of treatment in Quality of life during postoperative period, using the knee injury and osteoarthritis outcome score (KOOS)